CLINICAL TRIAL: NCT05049837
Title: PROSPECT - Profiling of Resistance Patterns & Oncogenic Signaling Pathways in Evaluation of Cancers of the Thorax and Therapeutic Target Identification
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LAB07-0233; 5R01CA157450-05 (NIH); 5R01CA183793 (NIH); 1R01CA205150-01 (NIH); NCI-2021-09810 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Cancer of Thorax
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Specific Aim 1: 600 cases: two normal and two tumor formalin-fixed tissue samples
  Interventions: Other: Group Specific Aim 1
- Specific Aim 2: 600 cases: two normal and two tumor formalin-fixed tissue samples.
  Interventions: Other: Group Specific Aim 2
- Specific Aim 3: 600 cases, including 150 patients who had received neoadjuvant therapy and 450 patients who had not. Two normal and two tumor formalin-fixed tissue samples.
  Interventions: Other: Group Specific Aim 3
- Specific Aim 4: 600 cases; including 150 patients who will receive neoadjuvant chemotherapy, 150 patients who received or will receive postoperative adjuvant chemotherapy, and 300 patients who did not receive or will not receive neoadjuvant or adjuvant chemotherapy. Two normal and two tumor formalin-fixed tissue samples
  Interventions: Other: Group Specific Aim 4
- Specific Aim 5: 600 cases; two normal and two tumor formalin-fixed tissue samples
  Interventions: Other: Group Specific Aim 5
- Specific Aim 6: 210 cases (of the 600 above), one normal and one tumor formalin-fixed histology sections obtained from formalin-fixed and paraffin- embedded tissue samples.
  Interventions: Other: Group Specific Aim 6

INTERVENTIONS:
Other: Group Specific Aim 1 — 600 cases: two normal and two tumor formalin-fixed tissue samples
  Groups: Specific Aim 1
Other: Group Specific Aim 2 — 600 cases: two normal and two tumor formalin-fixed tissue samples.
  Groups: Specific Aim 2
Other: Group Specific Aim 3 — 600 cases, including 150 patients who had received neoadjuvant therapy and 450 patients who had not. Two normal and two tumor formalin-fixed tissue samples
  Groups: Specific Aim 3
Other: Group Specific Aim 4 — 600 cases; including 150 patients who will receive neoadjuvant chemotherapy, 150 patients who received or will receive postoperative adjuvant chemotherapy, and 300 patients who did not receive or will not receive neoadjuvant or adjuvant chemotherapy. Two normal and two tumor formalin-fixed tissue samples
  Groups: Specific Aim 4
Other: Group Specific Aim 5 — 600 cases; two normal and two tumor formalin-fixed tissue samples
  Groups: Specific Aim 5
Other: Group Specific Aim 6 — 210 cases (of the 600 above), one normal and one tumor formalin-fixed histology sections obtained from formalin-fixed and paraffin- embedded tissue samples.
  Groups: Specific Aim 6

SUMMARY:
In this Project, we will use therapeutic target -focused (TTF) profiling, genome-wide mRNA profiling and assessments of tumor phosphopeptides and DNA that are shed into the blood stream to define how various molecular factors alone and in combination relate to resistance to therapy, to prognosis, and to metastatic patterns at relapse. We will examine how the presence of factors that drive cell growth, antagonize apoptosis, or confer resistance in other ways may counter the effect of systemic therapies and/or promote rapid tumor recurrence. In this way, we will identify new, previously unappreciated potential therapeutic targets while also identifying which targets are most likely to increase resistance to therapy and worsen prognosis.

DETAILED DESCRIPTION:
Objectives:

1. To develop a therapeutic target -focused (TTF) profiling platform and to use it in vitro to identify potential therapeutic targets associated with therapeutic resistance and to develop novel approaches against these potential targets.
2. To use tumor tissue TTF profiling along with genome wide mRNA profiling, serum phosphopeptide profiling and plasma DNA profiling to identify and evaluate molecular targets and pathways that contribute to therapeutic sensitivity or resistance, prognosis, and recurrence patterns in patients with operable non-small cell lung carcinoma (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

Eligible patients should be ones who have stage I-IIIA non-small cell lung cancer (NSCLC) and undergo surgical resection with or without neoadjuvant chemotherapy as part of standard treatment, and have a information of demographics, smoking history, preoperative clinical data, and follow -up data including adjuvant therapy, relapse, and treatment at relapse.

We will include the three major NSCLC histologic subtypes, adenocarcinoma, squamous cell carcinoma, and large cell carcinoma -

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center (Lung Cancer Patients)
  Patients should be ones who have stage I-IIIA non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 7200 (Estimated)
Dates: Start 2007-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop a therapeutic target -focused (TTF) profiling platform and to use it in vitro to identify potential therapeutic targets associated with therapeutic resistance and to develop novel approaches against these potential targets. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Luisa M Solis Soto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Caner Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org